CLINICAL TRIAL: NCT00401622
Title: Clinical Benefits of a Blood Glucose Monitoring System in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeScan (Industry)
Collaborators: Synexus(UK) (Unknown); CPS(UK) (Unknown); Battelle CRO(US) (Unknown); RPS CRO(US) (Unknown); Robertson Centre For Biostatistics (UK) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CR-1039797
Record Dates: First submitted 2006-11-16; First posted 2006-11-20 (Estimated); Results first posted 2010-09-16 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OneTouch® Ultra®2 system (Experimental): Test care group assigned to OneTouch® Ultra®2 system
  Interventions: Behavioral: OneTouch® Ultra®2 System
- Standard care (Active Comparator): Control group receiving standard care with a traditional blood glucose monitoring system
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: OneTouch® Ultra®2 System — Education and self-monitoring of blood glucose performed with OneTouch® Ultra®2 System that includes the Simple Start™ home-based education program
  Arms: OneTouch® Ultra®2 system
Behavioral: Standard care — Standard education and self-monitoring of blood glucose performed with traditional meter systems
  Arms: Standard care

SUMMARY:
Clinical benefits of the OneTouch® Ultra®2 BGMS versus standard BGMS during 52 weeks of use.

ELIGIBILITY:
Inclusion Criteria:·

* Current diagnosis of type 2 diabetes
* Diagnosed at least 3 months prior to the start of the study but not more than 15 years from the start of the study
* Stable regimen (i.e., no changes in therapeutic regimen) for the past three months
* Baseline HbA1c of 7.0 to 8.9%, inclusive

Exclusion Criteria:

* Using insulin
* Using oral agents that target post-prandial hyperglycemia (Note: These medications may be added during the study)
* Known history of anemia or disorders associated with anemia
* Has previously used the devices being tested in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2006-10-01 (Actual); Primary Completion 2009-01-01 (Actual); Study Completion 2009-01-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (10):
  - Phoenix, Arizona
  - San Diego, California
  - Wilmington, Delaware
  - Hollywood, Florida
  - Dawsonville, Georgia
  - Whitehouse Station, New Jersey
  - East Syracuse, New York
  - Endwell, New York
  - Syracuse, New York
  - San Antonio, Texas
- Canada (2):
  - Oshawa, Ontario
  - Windsor, Ontario
- United Kingdom (6):
  - Reading, Berkshire
  - Llanishen, Cardiff
  - Buckshaw Village, Chorley
  - Lloyd Street North, Manchester
  - Glasgow, Scotland
  - Claygate, Surrey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted at 18 study sites at various locations in the UK (6 Sites), US (10 Sites) and Canada (2 Sites). The first subject was enrolled on 10th October 2006 and the last Subject completed the study on 28th December 2008. Participating sites included family practice centres (US and UK) and hospital based clinical sites in the US.
Period: Overall Study
Arm/Group | OneTouch® Ultra®2 System | Standard Care
Started | 160 | 160
Completed | 126 | 117
Not Completed | 34 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OneTouch® Ultra®2 System | Standard Care | Total
Number analyzed (Participants) | 160 | 160 | 320
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 101 | 101 | 202
  >=65 years | 59 | 59 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (10.97) | 61.1 (10.54) | 60.8 (10.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 69 | 129
  Male | 100 | 91 | 191
Region of Enrollment [Number; unit: participants]
  United States | 109 | 103 | 212
  Canada | 12 | 9 | 21
  United Kingdom | 39 | 48 | 87
Baseline A1C [Mean (Standard Deviation); unit: Percentage] | 7.6 (0.48) | 7.6 (0.49) | 7.6 (0.49)
Fasting glucose [Mean (Standard Deviation); unit: mg/dl] | 141.1 (33.40) | 144.8 (39.19) | 143.0 (36.41)

OUTCOME MEASURES:

1. Secondary Outcome: Change in Daily Glycemic Excursions Between the OneTouch® Ultra®2 and Control BGMS.
Time Frame: 52 wks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | OneTouch® Ultra®2 System | Standard Care
Number analyzed (Participants) | 115 | 101
mg/dL | 102.7 (49.03) [-7.24 to 22.36] | 105.8 (38.17) [0 to 0]
Statistical Analysis 1: Comparison: OneTouch® Ultra®2 System vs Standard Care; Test type: Superiority or Other; p = 0.31, t-test, 2 sided; Mean Difference (Final Values) = 7.56, 95% CI 2-sided [-7.24 to 22.36], Standard Error of Mean 7.51

2. Primary Outcome: Change in A1C From Baseline to Week 52 Between the OneTouch® Ultra®2 and Control BGMS.
Time Frame: From baseline to 52 wks
Population: The study was designed to give 84% power to detect a 0.5% difference in the change of A1C between both groups
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | OneTouch® Ultra®2 System | Standard Care
Number analyzed (Participants) | 125 | 116
Percentage | -0.35 (0.073) [-0.38 to 0.04] | -0.18 (0.076) [0 to 0]
Statistical Analysis 1: Comparison: OneTouch® Ultra®2 System vs Standard Care; Change in A1C from baseline to week 52 between the OneTouch® Ultra®2 and control BGMS; Test type: Superiority or Other; p = 0.45, ANCOVA; Visit 1 A1c measurement used as the covariate; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.38 to 0.04], Standard Error of Mean 0.11

ADVERSE EVENTS:
Arm/Group | OneTouch® Ultra®2 System | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/160 | 1/160
Other Adverse Events (participants affected / at risk) | 0/160 | 0/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OneTouch® Ultra®2 System (N=160) | Standard Care (N=160)
BLOCKED ARTERIES ACROSS GROIN (Vascular disorders) | 0 (0) | 1 (1) — SUBJECT 36-019 03JUL2008 - 08 JUL 2008. Tx: BYPASS OPERATION REQUIRED IN-PATIENT HOSPITALIZATION SEVERE REMOTE CAUSALITY NOT A SADE RECOVERED

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days